CLINICAL TRIAL: NCT03357731
Title: A Multicenter, Randomized, Double-Blind, Placebo- and Active-Controlled, Cross-over Phase 2 Study of Continuous 5-Hour Intravenous Infusions of BMS-986231 in Patients With Heart Failure and Impaired Systolic Function
Brief Title: A Study of Continuous Infusions of HNO (Nitroxyl) Donor in Patients With Heart Failure and Impaired Systolic Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CV013-020; 2016-003586-26 (EudraCT Number)
Record Dates: First submitted 2017-10-31; First posted 2017-11-30 (Actual); Results first posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure; Cardiac Failure; Reduced Ventricular Ejection Fraction
MeSH Terms: conditions — Heart Failure | interventions — Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo/BMS-986231/NTG (Experimental): administered in a cross over design with 5-hour infusions and 5-28 day wash-out periods
  Interventions: Drug: HNO Donor; Drug: Nitroglycerin (NTG); Other: Placebo
- Placebo/NTG/BMS-986231 (Experimental): administered in a cross over design with 5-hour infusions and 5-28 day wash-out periods
  Interventions: Drug: HNO Donor; Drug: Nitroglycerin (NTG); Other: Placebo
- NTG/Placebo/BMS-986231 (Experimental): administered in a cross over design with 5-hour infusions and 5-28 day wash-out periods
  Interventions: Drug: HNO Donor; Drug: Nitroglycerin (NTG); Other: Placebo
- NTG/BMS-986231/Placebo (Experimental): administered in a cross over design with 5-hour infusions and 5-28 day wash-out periods
  Interventions: Drug: HNO Donor; Drug: Nitroglycerin (NTG); Other: Placebo
- BMS-986231/Placebo/NTG (Experimental): administered in a cross over design with 5-hour infusions and 5-28 day wash-out periods
  Interventions: Drug: HNO Donor; Drug: Nitroglycerin (NTG); Other: Placebo
- BMS-986231/NTG/Placebo (Experimental): administered in a cross over design with 5-hour infusions and 5-28 day wash-out periods
  Interventions: Drug: HNO Donor; Drug: Nitroglycerin (NTG); Other: Placebo

INTERVENTIONS:
Drug: HNO Donor — Infusion
  Other Names: BMS-986231
Drug: Nitroglycerin (NTG) — Infusion
Other: Placebo — Infusion

SUMMARY:
The purpose of this study is to evaluate the effects of BMS-986231 on systolic and diastolic parameters in patients with heart failure and low ejection fraction.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Heart failure with reduced ejection fraction (LVEF on echocardiogram of 40% or less)
* Stable guideline directed therapy for heart failure including oral diuretics, ACEi, ARBs, ARNi, MRAs, and β blockers as tolerated, with no dose changes of these medications in the past 2 weeks
* Have screening values of NT pro-BNP ≥ 125 pg/mL (15 pmol/L) or BNP ≥ 35 pg/mL (10 pmol/L)

Exclusion Criteria:

* Systolic blood pressure (SBP) < 110 mm Hg at screening or pre-randomization
* Heart rate < 50 beats per minute (bpm) or > 90 bpm at screening or pre-randomization
* Permanent Atrial Fibrillation, Atrial Flutter or having Atrial Fibrillation, Atrial Flutter
* Estimated glomerular filtration rate (eGFR) < 15 ml/min/1.73 m2
* Ventricular assist device or prior heart transplant
* Prior solid organ transplant
* Body weight < 45 kg or ≥ 140 kg
* Low quality echocardiographic visualization windows and image acquisition
* Permanent paced rhythm (VVI, DDD or BiV pacing)

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (6):
  - Orange County Research Center, Tustin, California
  - Northwestern Medicine, Chicago, Illinois
  - Indiana University School of Medicine-Indianapolis, Indianapolis, Indiana
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Duke Advanced Heart and Lung Failure Clinic, Durham, North Carolina
  - Inova Heart and Vascular Institute, Falls Church, Virginia
- Japan (3):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Kawasaki, Kanagawa
  - Local Institution, Suita-shi, Osaka
- Local Institution, Groiningen, Netherlands
- United Kingdom (4):
  - Local Institution, Edinburgh
  - Local Institution, Glasgow
  - Local Institution, Harrow
  - Local Institution, London

REFERENCES:
- [Derived] Felker GM, Borentain M, Cleland JG, DeSouza MM, Kessler PD, O'Connor CM, Seiffert D, Teerlink JR, Voors AA, McMurray JJV. Rationale and design for the development of a novel nitroxyl donor in patients with acute heart failure. Eur J Heart Fail. 2019 Aug;21(8):1022-1031. doi: 10.1002/ejhf.1504. Epub 2019 Jun 6. PMID 31168885
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 49 participants assigned to treatment and 45 treated. Reasons not treated: 2 re-randomized; 1 randomized in error, screen failure; 1 no longer met study criteria.
  Note: Study designed for all participants to enter all 3 arms (reassignment of arms occurs every period change).
Groups:
- Sequence 1: Participants crossed-over from one therapy to the next following Day 1 treatment and a minimum 5-day washout period.
  3 treatments were given via 1 of 6 different order sequences across 3 total treatment periods, 1 treatment per period. Treatments were as follows: Placebo (PBO) BMS-986231 (drug) Nitroglycerin (NTG)
  Sequence of treatment for this group is as follows: PBO-drug-NTG
- Sequence 2: Participants crossed-over from one therapy to the next following Day 1 treatment and a minimum 5-day washout period.
  3 treatments were given via 1 of 6 different order sequences across 3 total treatment periods, 1 treatment per period. Treatments were as follows: Placebo (PBO) BMS-986231 (drug) Nitroglycerin (NTG)
  Sequence of treatment for this group is as follows: PBO-NTG-drug
- Sequence 3: Participants crossed-over from one therapy to the next following Day 1 treatment and a minimum 5-day washout period.
  3 treatments were given via 1 of 6 different order sequences across 3 total treatment periods, 1 treatment per period. Treatments were as follows: Placebo (PBO) BMS-986231 (drug) Nitroglycerin (NTG)
  Sequence of treatment for this group is as follows: NTG-PBO-drug
- Sequence 4: Participants crossed-over from one therapy to the next following Day 1 treatment and a minimum 5-day washout period.
  3 treatments were given via 1 of 6 different order sequences across 3 total treatment periods, 1 treatment per period. Treatments were as follows: Placebo (PBO) BMS-986231 (drug) Nitroglycerin (NTG)
  Sequence of treatment for this group is as follows: NTG-drug-PBO
- Sequence 5: Participants crossed-over from one therapy to the next following Day 1 treatment and a minimum 5-day washout period.
  3 treatments were given via 1 of 6 different order sequences across 3 total treatment periods, 1 treatment per period. Treatments were as follows: Placebo (PBO) BMS-986231 (drug) Nitroglycerin (NTG)
  Sequence of treatment for this group is as follows: drug-PBO-NTG
- Sequence 6: Participants crossed-over from one therapy to the next following Day 1 treatment and a minimum 5-day washout period.
  3 treatments were given via 1 of 6 different order sequences across 3 total treatment periods, 1 treatment per period. Treatments were as follows: Placebo (PBO) BMS-986231 (drug) Nitroglycerin (NTG)
  Sequence of treatment for this group is as follows: drug-NTG-PBO
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started (started = received Period 1 assigned treatment) | 8 | 7 | 7 | 7 | 8 | 8
Completed Period 1 (P1) | 8 (1 withdrew post-P1 completion/prior to P2 therapy due to acute cholecystitis, but returned for P2/P3) | 7 | 7 | 6 (1 discontinued P1 due to acute bradycardia and hypotension) | 7 (1 discontinued P1 due to hypotension but resumed P2/P3) | 8
Completed Period 2 (P2) | 8 | 7 | 7 | 4 (1 completed P1, did not proceed to P2/P3 (lost to follow-up); 1 discontinued P2 due to hypotension) | 7 (1 only completed P1, did not continue to P2/P3 (withdrew consent due to personal reasons)) | 7 (1 discontinued P2 due to an Adverse Event (AE))
Completed (completed = finished Period 3 (P3) assigned treatment) | 8 | 7 | 6 (1 discontinuation due to hypotension) | 4 | 7 | 7
Not Completed | 0 | 0 | 1 | 3 | 1 | 1
Not completed — Withdrew consent due to personal reasons | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Acute bradycardia and hypotension | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Hypotension | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Participants: Inclusive of all treatments, all periods. Note: Participants crossed-over from either placebo, drug or NTG arm to the next (in various sequence) following Day 1 treatment and a minimum 5-day washout period, per arm.
Arm/Group | Overall Participants
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (12.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 40
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Stroke Volume Index (SVI) Derived From the Velocity Time Integral at the Left Ventricular Outflow Tract (LVOT VTI) at the End of the 5-hour Infusion of BMS-986231, Versus Placebo
Description: The objective is to evaluate the effects of BMS-986231 on the left ventricular (LV) systolic function by stroke volume index (SVI) assessed by echocardiography compared to placebo.
Time Frame: at the end of the 5-hour infusion
Population: Intent to Treat (ITT) population: All randomized participants who started study drug infusion in at least one treatment period.
Measure: Mean (Standard Deviation); unit: mL/m^2
Groups:
- Placebo (PBO): Placebo-matching treatment. Note: Participants crossed-over from one arm to the next following Day 1 treatment and a minimum 5-day washout period, per arm.
  Treatment was given via 1 of 6 different order sequences across 3 total treatment periods. Participant therapy sequence assignment varies as follows:
  PBO-drug-NTG, PBO-NTG-drug, NTG-PBO-drug, NTG-drug-PBO, drug-PBO-NTG, drug-NTG-PBO
- BMS-986231: BMS-986231: 3 μg/kg/min for 10 min, followed by 6 μg/kg/min for 10 min, followed by 12 μg/kg/min for the rest of the 5-hour infusion.
  Note: Participants crossed-over from one arm to the next following Day 1 treatment and a minimum 5-day washout period, per arm.
  Treatment was given via 1 of 6 different order sequences across 3 total treatment periods. Participant therapy sequence assignment varies as follows:
  PBO-drug-NTG, PBO-NTG-drug, NTG-PBO-drug, NTG-drug-PBO, drug-PBO-NTG, drug-NTG-PBO
- Nitroglycerin (NTG): NTG: 20 μg/min for 10 min, followed by 40 μg/min for 10 min, followed by 80 μg/min for the rest of the 5-hour infusion Note: Participants crossed-over from one arm to the next following Day 1 treatment and a minimum 5-day washout period, per arm.
  Treatment was given via 1 of 6 different order sequences across 3 total treatment periods. Participant therapy sequence assignment varies as follows:
  PBO-drug-NTG, PBO-NTG-drug, NTG-PBO-drug, NTG-drug-PBO, drug-PBO-NTG, drug-NTG-PBO
Arm/Group | Placebo (PBO) | BMS-986231 | Nitroglycerin (NTG)
Number analyzed (Participants) | 39 | 37 | 0
mL/m^2 | 29.545 (7.0243) | 28.721 (9.0174) |
Statistical Analysis 1: Comparison: Placebo (PBO) vs BMS-986231; Test type: Superiority; p = 0.027, Kenward-Roger degree of freedom; Kenward-Roger degree of freedom is used to adjust the standard error of treatment effect; Mean Difference (Net) = -2.150, 95% CI 2-sided [-4.0432 to -0.2570], Standard Error of Mean 0.9242 — The modelled mean difference uses treatment sequence and difference of baselines as a covariates of the treatment effect

2. Secondary Outcome: Mean SVI Derived From LVOT VTI at the End of the 5-hour Infusion of BMS-986231, Versus NTG
Description: The objective is to evaluate the effects of BMS-986231 on the left ventricular (LV) systolic function by stroke volume index (SVI) assessed by echocardiography compared to NTG.
Time Frame: at the end of the 5-hour infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Placebo (PBO) | BMS-986231 | Nitroglycerin (NTG)
Number analyzed (Participants) | 0 | 37 | 41
mL/m^2 |  | 28.721 (9.0174) | 27.811 (7.9712)
Statistical Analysis 1: Comparison: BMS-986231 vs Nitroglycerin (NTG); Test type: Superiority; p = 0.846, Kenward-Roger degree of freedom; Kenward-Roger degree of freedom is used to adjust the standard error of treatment effect; Mean Difference (Net) = 0.193, 95% CI 2-sided [-1.8176 to 2.2042], Standard Error of Mean 0.9832 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Mean LVEF, Computed by Simpson's Method at the End of the 5-hour Infusion of BMS-986231, Versus Placebo and NTG
Description: Evaluate the effects of BMS-986231 on selected other left ventricular systolic and diastolic indices compared to placebo and NTG:
  LV ejection fraction
Time Frame: at the end of the 5-hour infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of blood pumped from the LV
Arm/Group | Placebo (PBO) | BMS-986231 | Nitroglycerin (NTG)
Number analyzed (Participants) | 38 | 36 | 42
Percentage of blood pumped from the LV | 31.9 (7.15) | 32.8 (8.24) | 33.5 (7.33)
Statistical Analysis 1: Comparison: Placebo (PBO) vs BMS-986231; Test type: Superiority; p = 0.177, Kenward-Roger degree of freedom; Kenward-Roger degree of freedom is used to adjust the standard error of treatment effect; Mean Difference (Net) = 1.3, 95% CI 2-sided [-0.62 to 3.19], Standard Error of Mean 0.93 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BMS-986231 vs Nitroglycerin (NTG); Test type: Superiority; p = 0.839, Kenward-Roger degree of freedom; Kenward-Roger degree of freedom is used to adjust the standard error of treatment effect; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.08 to 0.88], Standard Error of Mean 0.48 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Mean Cardiac Power Index at the End of the 5-hour Infusion of BMS-986231, Versus Placebo and NTG
Description: Evaluate the effects of BMS-986231 on selected other left ventricular systolic and diastolic indices compared to placebo and NTG:
  Mean LV power index
Time Frame: at the end of the 5-hour infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: watts per square meter (W/m^2)
Arm/Group | Placebo (PBO) | BMS-986231 | Nitroglycerin (NTG)
Number analyzed (Participants) | 35 | 36 | 39
watts per square meter (W/m^2) | 0.4122 (0.14404) | 0.3427 (0.10463) | 0.3568 (0.09184)
Statistical Analysis 1: Comparison: Placebo (PBO) vs BMS-986231; Test type: Superiority; p = 0.007, Kenward-Roger degree of freedom; Kenward-Roger degree of freedom is used to adjust the standard error of treatment effect; Mean Difference (Net) = -0.0977, 95% CI 2-sided [-0.16634 to -0.02915], Standard Error of Mean 0.03308 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BMS-986231 vs Nitroglycerin (NTG); Test type: Superiority; p = 0.103, Kenward-Roger degree of freedom; Kenward-Roger degree of freedom is used to adjust the standard error of treatment effect; Mean Difference (Net) = -0.0371, 95% CI 2-sided [-0.08243 to 0.00814], Standard Error of Mean 0.02194 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Mean Diastolic Indices: E/A and E/e' Ratio at the End of the 5-hour Infusion of BMS-986231, Versus Placebo and NTG
Description: Evaluate the effects of BMS-986231 on selected other left ventricular systolic and diastolic indices compared to placebo and NTG:
  Diastolic function
Time Frame: at the end of the 5-hour infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo (PBO) | BMS-986231 | Nitroglycerin (NTG)
Number analyzed (Participants) | 37 | 34 | 40
Ratio
  E/A ratio: number analyzed (Participants) | 36 | 31 | 36
  E/A ratio | 0.80 (0.278) | 0.73 (0.270) | 0.71 (0.310)
  E/e' ratio: number analyzed (Participants) | 35 | 32 | 37
  E/e' ratio | 9.42 (4.102) | 7.00 (2.464) | 7.81 (2.652)
Statistical Analysis 1: Comparison: Placebo (PBO) vs BMS-986231; E/A ratio; Test type: Superiority; p = 0.003, Kenward-Roger degree of freedom; Kenward-Roger degree of freedom is used to adjust the standard error of treatment effect; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.205 to -0.051], Standard Error of Mean 0.037 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BMS-986231 vs Nitroglycerin (NTG); E/A ratio; Test type: Superiority; p = 0.904, Kenward-Roger degree of freedom; Kenward-Roger degree of freedom is used to adjust the standard error of treatment effect; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.051 to 0.057], Standard Error of Mean 0.026 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo (PBO) vs BMS-986231; E/e' ratio; Test type: Superiority; p = 0.006, Kenward-Roger degree of freedom; Kenward-Roger degree of freedom is used to adjust the standard error of treatment effect; Mean Difference (Net) = -1.66, 95% CI 2-sided [-2.763 to -0.549], Standard Error of Mean 0.527 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: BMS-986231 vs Nitroglycerin (NTG); E/e' ratio; Test type: Superiority; p = 0.503, Kenward-Roger degree of freedom; Kenward-Roger degree of freedom is used to adjust the standard error of treatment effect; Mean Difference (Net) = -0.27, 95% CI 2-sided [-1.085 to 0.550], Standard Error of Mean 0.392 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Mean Diastolic Indices: Annular e' Velocity at the End of the 5-hour Infusion of BMS-986231, Versus Placebo and NTG
Description: as for outcome 5
Time Frame: at the end of the 5-hour infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Placebo (PBO) | BMS-986231 | Nitroglycerin (NTG)
Number analyzed (Participants) | 37 | 34 | 40
cm/sec | 7.18 (2.467) | 8.07 (2.333) | 7.18 (2.143)
Statistical Analysis 1: Comparison: Placebo (PBO) vs BMS-986231; annular e' velocity; Test type: Superiority; p = 0.994, Kenward-Roger degree of freedom; Kenward-Roger degree of freedom is used to adjust the standard error of treatment effect; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.827 to 0.820], Standard Error of Mean 0.398 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BMS-986231 vs Nitroglycerin (NTG); annular e' velocity; Test type: Superiority; p = 0.073, Kenward-Roger degree of freedom; Kenward-Roger degree of freedom is used to adjust the standard error of treatment effect; Mean Difference (Net) = 0.48, 95% CI 2-sided [-0.049 to 1.013], Standard Error of Mean 0.258 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Mean LV Global Longitudinal Strain, Computed Using STE at the End of the 5-hour Infusion of BMS-986231, Versus Placebo and NTG
Description: Evaluate the effects of BMS-986231 on selected other left ventricular systolic and diastolic indices compared to placebo and NTG:
  LV global longitudinal strain
Time Frame: at the end of the 5-hour infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of blood pumped from the LV
Arm/Group | Placebo (PBO) | BMS-986231 | Nitroglycerin (NTG)
Number analyzed (Participants) | 38 | 36 | 43
Percentage of blood pumped from the LV | -11.98 (2.860) | -11.94 (3.458) | -11.36 (3.067)
Statistical Analysis 1: Comparison: Placebo (PBO) vs BMS-986231; Test type: Superiority; p = 0.705, Kenward-Roger degree of freedom; Kenward-Roger degree of freedom is used to adjust the standard error of treatment effect; Mean Difference (Net) = 0.15, 95% CI 2-sided [-0.670 to 0.976], Standard Error of Mean 0.400 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BMS-986231 vs Nitroglycerin (NTG); Test type: Superiority; p = 0.105, Kenward-Roger degree of freedom; Kenward-Roger degree of freedom is used to adjust the standard error of treatment effect; Mean Difference (Net) = -0.68, 95% CI 2-sided [-1.504 to 0.151], Standard Error of Mean 0.404 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first dose to 30 days post last dose (approximately 3 months)
Arm/Group | Placebo (PBO) | BMS-986231 | Nitroglycerin (NTG)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/42 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/42 | 1/44
Other Adverse Events (participants affected / at risk) | 2/40 | 12/42 | 10/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (PBO) (N=40) | BMS-986231 (N=42) | Nitroglycerin (NTG) (N=44)
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (PBO) (N=40) | BMS-986231 (N=42) | Nitroglycerin (NTG) (N=44)
Headache (Nervous system disorders) | 2 | 10 | 7
Hypotension (Vascular disorders) | 0 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT03357731/SAP_000.pdf
  • Study Protocol (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT03357731/Prot_001.pdf